CLINICAL TRIAL: NCT03392194
Title: Adapting Sleep and Yoga Interventions for Maximal Effectiveness in Low Income Populations
Acronym: CALYPSO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Susan Redline, Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P002349; 1R34AT008923-01 (NIH)
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Results first posted 2019-08-21 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Sleep
Keywords: Behavioral interventions; Sleep hygiene; Yoga; Community research; Short sleep duration; Low-income population
MeSH Terms: conditions — Sleep Hygiene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep hygiene & Yoga (SH+Y) (Experimental): Participants will receive the sleep hygiene intervention, which includes 2 sleep hygiene sessions and 10 weeks of maintenance assessment. After completing the SH sessions, they will receive 10 weeks of the yoga intervention (8 in-person yoga sessions and 2 weeks of yoga home practice maintenance assessment).
  Interventions: Behavioral: Sleep hygiene intervention; Behavioral: Yoga intervention
- Sleep hygiene (SH) (Active Comparator): Participants will receive the sleep hygiene intervention, which includes 2 sleep hygiene sessions and 10 weeks of maintenance assessment.
  Interventions: Behavioral: Sleep hygiene intervention

INTERVENTIONS:
Behavioral: Sleep hygiene intervention — The community-adapted SH intervention includes 2 group sessions. (1) teach the importance of sleep and the core components of SH; distribute and explain the daily sleep log (2) facilitate an open discussion where participants share challenges and experiences implementing a SH goal.
Behavioral: Yoga intervention — Following the SH intervention, participants randomized to the SH+Y arm will participate in 8 weekly beginner level yoga classes. Classes will increase participants' skill and comfort with yoga postures and relaxing breathing exercises so that participants can adopt an evening yoga practice (10 weeks).
  Arms: Sleep hygiene & Yoga (SH+Y)

SUMMARY:
The purpose of this study is to evaluate the feasibility of conducting a future randomized control trial that will compare the efficacy of sleep behavioral interventions in a high-risk community including adapted sleep hygiene and yoga. The investigators will conduct a 40 person 12-week randomized control trial (RCT) in low-income housing population where half the participants will receive a community adapted sleep hygiene intervention (SH) and half will receive a community adapted sleep hygiene intervention and a yoga intervention. The investigators will evaluate the feasibility of recruiting from our target community, randomizing individuals to interventions delivered in community rooms with home-based practices, and delivering the targeted interventions with high adherence and fidelity.

DETAILED DESCRIPTION:
Inadequate sleep is highly prevalent in low-socioeconomic status (SES) and minority groups and associated with multiple health problems. The root causes of inadequate sleep are often related to behavioral practices and stress, both of which may be favorably impacted using socio-contextually appropriate sleep hygiene recommendations and mind-body practices such as yoga. A preliminary RCT that will address the role of sleep behavioral interventions in a high-risk community will be conducted. This evidence is needed to guide mind-body therapies in low-SES communities in which such strategies are under-utilized to improve health.

The investigators have assembled a multidisciplinary team of experts in sleep medicine, complementary and integrative health, behavioral medicine, community engagement, social epidemiology, and clinical trials to conduct a planning study to adapt behavioral sleep interventions for residents in urban low-income housing and to evaluate their uptake and fidelity. The investigators have conducted qualitative formative evaluation work and conducted modified SH and Yoga pilot studies. In this phase, the investigators will deliver a 12-week trial testing the feasibility of (1) an adapted sleep hygiene intervention (SH) and (2) yoga + adapted sleep hygiene intervention SH+Y):

A. A Sleep Hygiene (SH) Intervention, addressing: beliefs and attitudes towards sleep; challenges for adhering to sleep hygiene recommendations given chaotic family routines, work schedules and bedroom conditions; strategies for overcoming barriers, and prioritization of recommendations most likely to be efficacious.

B. A Yoga (Y) Intervention: intervention intensity/duration and class format; tailored home-based recommendations for bedtime practice combining meditation, breathing and postures; tools to assess and enhance adherence; race/ethnicity concordance of the instructor and student; and use of peer yoga assistants.

The investigators aim to conduct a 40 person 12-week RCT of SH vs SH+Y to inform the design of a future large-scale RCT. The investigators will evaluate the feasibility of recruiting from our target community, randomizing individuals to interventions delivered in community rooms with home-based practices, and delivering the targeted interventions with high adherence and fidelity. The following will be evaluated:

* Reach of the target population: The number of potentially eligible individuals approached to participate will be tracked as well as the characteristics of individuals who do and do not choose to participate, and differences will be assessed. Reasons for choosing not to participate will be assessed using open ended questions (e.g., burden, perception of yoga, needs, etc.).
* Adoption and adherence: the proportion of individuals that sustain participation throughout the intervention will be assessed, and quantify attendance at classes and home-practices through logs and interim phone interviews. The investigators will describe patterns of dropout rates and adherence to the interventions by key demographic factors and by moderating and mediating factors.
* Implementation-consistency of delivery of the intervention: a checklist of core intervention elements will be used to document the degree to which core elements of the intervention was delivered as specified in the protocol.

The investigators will also assess the feasibility of collecting a range of baseline, outcome, process and mediator data and to generate data to support use of specific measures in a later trial, including patterns of missingness of data, distributions of data, correlations between outcomes, baseline factors and mediators, and evaluation of "dose-response" associations between time in intervention and sleep duration and efficiency.

Power analysis (sample size, evaluable subjects, etc.): The study is designed for feasibility and not powered to test the intervention effect. The SH+Y intervention will be considered as potentially efficacious if the estimates for the change scores (post-pre within and between group changes and their 95% confidence intervals) are consistent with clinically significant improvements in sleep duration (actigraphy sleep increases by > 30 minutes), sleep quality improves by > 0.3 standard deviations), or sleep hygiene (reduction in deviation in wake time relative to recommended wake time > 25%). The investigators will consider inclusion of specific measurements (mediators) in a future RCT based on: <10% missingness; correlation of change score or baseline score with outcomes of >.20; absence of redundancy with a simpler metric (r<.80).

ELIGIBILITY:
Inclusion Criteria:

* Verbally proficient in English
* Self-reported average (over the prior month) weekday sleep duration of < 6 hours
* Reside in a public housing

Exclusion Criteria:

* Severe physical conditions preventing participation in yoga, including major surgery or head injury in the prior 3 months, or unstable vertebral injury with inability to sit or lie down for 5 or more minutes; or glaucoma
* Major psychiatric disease (e.g. schizophrenia, depression, PTSD) resulting in hospitalization in the last year; or disease severity that, in the opinion of the investigator, would make it difficult for the participant to partake in the study activities.
* Severe sleep disorders: self-report of physician diagnosed insomnia requiring hypnotics more than 3 times/ week or an untreated known sleep disorder (sleep apnea, RLS), that in the opinion of the investigator, would make it difficult for the participant to achieve sleep hygiene goals.
* Needing an assistive device such as a walker or cane, frequent falls, history of stroke resulting in weakness or numbness interfering with moving easily, or other problems causing ongoing balance issues and difficulty walking
* Yoga class participation in last 6 weeks
* Known pregnancy.
* Participation in prior sleep and yoga study pilots

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Redline, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spadola CE, Rottapel R, Khandpur N, Kontos E, Bertisch SM, Johnson DA, Quante M, Khalsa SBS, Saper RB, Redline S. Enhancing yoga participation: A qualitative investigation of barriers and facilitators to yoga among predominantly racial/ethnic minority, low-income adults. Complement Ther Clin Pract. 2017 Nov;29:97-104. doi: 10.1016/j.ctcp.2017.09.001. Epub 2017 Sep 4. PMID 29122272

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January-March 2018, participants were recruited from two affordable housing communities. Convenience and snowball sampling methods were employed. Study staff and community partners provided information to interested participants at community events and distributed flyers and postcards throughout the communities.
Pre-assignment Details: Sleep hygiene (SH) group sessions served as a run-in period for randomization. Participants were consented to participate in the research study (n=38) and then attended two SH group session. At the end of the second SH session, participants were randomized to the SH-arm or the sleep hygiene and yoga (SH+Y) arm (n=33).
Period: Overall Study
Arm/Group | Sleep Hygiene & Yoga (SH+Y) | Sleep Hygiene (SH)
Started | 16 | 17
Completed | 14 | 15
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Conflicts with personal schedule | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline population includes those who consented to participate in the study and were randomized to the SH arm or SH+Y arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sleep Hygiene & Yoga (SH+Y) | Sleep Hygiene (SH) | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 29
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.44 (14.74) | 47.29 (10.83) | 45.91 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 10 | 9 | 19
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 3 | 2 | 5
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 3 | 2 | 5
Sleep Duration [Mean (Standard Deviation); unit: minutes/night] — Population: The number analyzed in rows differs from overall due to missing count (not all participants were compliant or successful in wearing actigraphy)
  minutes/night
    number analyzed (Participants) | 15 | 15 | 30
    (all) | 400.69 (75.45) | 418.06 (66.07) | 409.37 (70.24)

OUTCOME MEASURES:

1. Primary Outcome: Sleep Duration
Description: Change in sleep duration from baseline to follow-up measure by actigraphs. We will conduct a repeated measures ANCOVA, modeling time, intervention group and a time*intervention interaction. We will explore change in stress, anxiety, depressive symptoms, mindfulness, and sleep hygiene score as potential explanatory variables.
Time Frame: 12 weeks
Population: The missing count is based on 21 participants having adequate quality actigraphy data at both baseline and endpoint
Measure: Mean (Standard Deviation); unit: minutes/night
Arm/Group | Sleep Hygiene & Yoga (SH+Y) | Sleep Hygiene (SH)
Number analyzed (Participants) | 11 | 14
minutes/night | -0.91 (43.87) | -2.93 (66.92)
Statistical Analysis 1: Comparison: Sleep Hygiene & Yoga (SH+Y) vs Sleep Hygiene (SH); Null hypothesis: There is no difference in change in sleep duration between the two intervention arms; Test type: Other — The purpose of this small pilot randomized control trial (RCT) was to assess feasibility and acceptability of conducting community based sleep hygiene and yoga interventions, to be scaled and tested in a future, larger RCT; p = 0.932, t-test, 2 sided; Due to main findings, analysis to explore potential mediators of effect were not pursued, despite original plan to explore explanatory variables; Mean Difference (Net) = -2.02, 95% CI 2-sided [-46.35 to 50.39]

ADVERSE EVENTS:
Time Frame: Five months.
Arm/Group | Sleep Hygiene & Yoga (SH+Y) | Sleep Hygiene (SH)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17
Other Adverse Events (participants affected / at risk) | 8/16 | 6/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sleep Hygiene & Yoga (SH+Y) (N=16) | Sleep Hygiene (SH) (N=17)
Cellulitis (foot) (Infections and infestations) | 0 (0) | 1 (2) — Participant reported inflammation in foot. When to ER and was prescribed antibiotics (Clindamycin) for cellulitis. Participant had a follow-up visit with primary care provider.
Mild rash (actigraph) (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) — Participants reported mild rash or irritation on wrist from wearing actigraph watch.
Ear infection (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Back pain/spasm (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) — short-term back or shoulder pain or spasm
Leg pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Root canal infection (Infections and infestations) | 1 (1) | 0 (0) — Participant had a root canal followed by infection; received treatment.
Arm and chest pain (Cardiac disorders) | 2 (2) | 0 (0) — Pain in arm, chest, or heart leading to emergency department visit.
Scratched cornea (Eye disorders) | 0 (0) | 1 (1) — Scratched cornea and received antibiotics treatment
Infection (Infections and infestations) | 0 (0) | 1 (2) — Reported abdominal abscess and associated infection; was actively seeking medical treatment.

LIMITATIONS AND CAVEATS:
This study was a developmental pilot to test novel interventions in the community. At this stage, sample sizes were not developed to achieve power and statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT03392194/Prot_SAP_002.pdf
  • Informed Consent Form (2018-04-11): https://cdn.clinicaltrials.gov/large-docs/94/NCT03392194/ICF_003.pdf